CLINICAL TRIAL: NCT02198092
Title: Preliminary Evaluation of Septin9 in Patients With Hereditary Colon Cancer Syndromes
Acronym: Septin9
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Epigenomics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 816593
Record Dates: First submitted 2014-07-15; First posted 2014-07-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Familial Adenomatous Polyposis; Map Syndrome; Lynch Syndrome; Hnpcc; Colorectal Cancer
Keywords: familial adenomatous polyposis; multiple adenomatous polyposis; lynch syndrome; hnpcc; colorectal cancer; genetic syndrome; epigenomics; septin9
MeSH Terms: conditions — Adenomatous Polyposis Coli; Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be used as per the study protocol. Consented subjects will provide at least 10 ml but not more than 20 ml (for repeating testing) of blood at each time point for Epi proColon testing. An additional volume of up to 10 ml anticoagulated blood will be drawn for circulating colonic epithelial cell analysis at each time point. Blood samples will be stored and will only be used in future research with the express written permission of study subjects. Subjects may withdraw consent from the study or for future use of blood samples at any time.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patient Group FAP: Clinical diagnosis of familial adenomatous polyposis (FAP).
  The patients of the disease and control groups participating in the study are followed up clinically and with blood draws at least every 6 months for the duration of 2 years. These follow-ups might be more frequent, if warranted by the clinical course of the individual disease in the participating patients. Blood draws in FAP patients should always be accompanied by blood draws in their family member controls.
  If colectomy is performed in a patient of any disease group within the study participation period, additional blood draws will occur prior to any surgical bowel preparation and within a 28-day window after surgery.
  Interventions: Other: Epi proColon Testing
- Patient Group Lynch Syndrome: Clinical diagnosis of Lynch Syndrome, also known as HNPCC.
  The patients of the disease and control groups participating in the study are followed up clinically and with blood draws at least every 6 months for the duration of 2 years. These follow-ups might be more frequent, if warranted by the clinical course of the individual disease in the participating patients.
  If colectomy is performed in a patient of any disease group within the study participation period, additional blood draws will occur prior to any surgical bowel preparation and within a 28-day window after surgery.
  Interventions: Other: Epi proColon Testing
- Patient Group MAP / MYH: Clinical diagnosis of MYH-associated polyposis and presence of more than 20 colon polyps.
  The patients of the disease and control groups participating in the study are followed up clinically and with blood draws at least every 6 months for the duration of 2 years. The follow-ups might be more frequent, if warranted by the clinical course of the individual disease in the participating patients.
  If colectomy is performed in a patient of any disease group within the study participation period, additional blood draws will occur prior to any surgical bowel preparation and within a 28-day window after surgery.
  Interventions: Other: Epi proColon Testing
- Control Group (FAP Genetically-Related): Genetically related family member of enrolled FAP patient.
  Controls, i.e. relatives of patients: Willingness to give blood at each routine follow-up as advised for the diseased relative.
  The patients of the control group participating in the study are followed up clinically and with blood draws at least every 6 months for the duration of 2 years. These follow-ups might be more frequent, if warranted by the clinical course of the individual disease in the participating FAP patients.
  If colectomy is performed in a FAP patient of any disease group within the study participation period, additional blood draws will occur prior to any surgical bowel preparation and within a 28-day window after surgery.
  Blood draws in FAP patients should always be accompanied by blood draws in their family member controls.
  Interventions: Other: Epi proColon Testing

INTERVENTIONS:
Other: Epi proColon Testing — Plasma specimens will be collected and processed according to the Instructions for Use of the Epi proColon investigational device.
  For circulating colonic epithelial cell analysis, at least one ml whole blood will be required for analysis. Samples will be analyzed for circulating epithelial cells using the geometrically enhanced immunocapture device (GEDI; Gleghorn et al., 2009). Circulating epithelial cells will be captured using EpCAM antibodies and quantified by immunofluorescence microscopy as defined as cells that are DAPI+, CK+, CD45-. Captured cells will be fixed and stored at -20˚C.

SUMMARY:
This is an observational, case-control study evaluating the quantitative level of Septin9 in plasma pre- and post-colectomy in hereditary colorectal cancer (CRC) syndrome patients (Familial Adenomatous Polyposis (FAP), Lynch syndrome (also known as HNPCC), and Multiple Adenomatous Polyposis (MAP, also known as MYK/MYH) cases) and genetically related FAP-family members as controls and references.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided
* Age > or = to 18 years of age
* Patient group FAP

  - Clinical diagnosis of familial adenomatous polyposis
* Patient group Lynch syndrome Clinical diagnosis of Lynch syndrome
* Patient group MAP

  - Clinical diagnosis of MYH-associated polyposis and presence of more than 20 colon polyps
* Control group (FAP)

  - Genetically related family member of patient
* Patients: Able and willing to attend routine follow-up as advised
* Controls, i.e. relatives of patients: Willingness to give blood at each routine follow-up as advised for the diseased relative

Exclusion Criteria:

* Known infection with Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV)
* Current diagnosis of colorectal cancer
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age > or = to 18 years of age Clinical diagnosis of familial adenomatous polyposis Clinical diagnosis of Lynch syndrome Clinical diagnosis of MYH-associated polyposis and presence of more than 20 colon polyps Genetically related family member of patients with clinical diagnosis of FAP for Control group
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Septin9 Plasma Levels | Up to 2 years
  The primary objective of the study is the observational analysis of quantitative Septin9 plasma levels over time in hereditary CRC syndrome patients pre- and post-colectomy.

SECONDARY OUTCOMES:
Septin9 Plasma Levels Versus Polyps | Up to 2 years
  • Correlation of quantitative Septin9 plasma levels with the approx. number of polyps
Pre- and Post-Colectomy Colonic Epithelial Cell Numbers | Up to 2 years
  • Correlation of circulating colonic epithelial cell number pre- and post-colectomy
Septin9 Levels Versus Circulating Colonic Epithelial Cell Numbers | Up to 2 years
  • Correlation of circulating colonic epithelial cell number with Septin9 levels

OTHER OUTCOMES:
Septin9 Monitoring in Individual Groups | Up to 2 years
  The primary endpoint of the study is the completion of Septin9 monitoring in the individual patient disease groups (or family controls) over a period of two years or in case of colectomy within 28 days after colectomy. The endpoint is defined as the documented receipt of blood draws at least every six months on the scheduled healthcare visit at the institute after enrollment over the two years participation period. If any patient needs to undergo colectomy within the two years of study participation, the endpoint is defined as documented receipt of both blood draws occured prior to any surgical bowel preparation and 28 days at the latest after surgery.
Circulating Colonic Epithelial Cells at Blood Draws | Up to 2 years
  The secondary endpoints of the study are the documented results of the circulating colonic epithelial cell numbers for each blood draw performed.

CONTACTS AND LOCATIONS:
Overall Officials: Bryson Katona, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Rustgi AK. The genetics of hereditary colon cancer. Genes Dev. 2007 Oct 15;21(20):2525-38. doi: 10.1101/gad.1593107. PMID 17938238
- [Background] Galiatsatos P, Foulkes WD. Familial adenomatous polyposis. Am J Gastroenterol. 2006 Feb;101(2):385-98. doi: 10.1111/j.1572-0241.2006.00375.x. PMID 16454848
- [Background] Lofton-Day C, Model F, Devos T, Tetzner R, Distler J, Schuster M, Song X, Lesche R, Liebenberg V, Ebert M, Molnar B, Grutzmann R, Pilarsky C, Sledziewski A. DNA methylation biomarkers for blood-based colorectal cancer screening. Clin Chem. 2008 Feb;54(2):414-23. doi: 10.1373/clinchem.2007.095992. Epub 2007 Dec 18. PMID 18089654